CLINICAL TRIAL: NCT00905762
Title: A Single-Center, Randomized, Masked Study Comparing the Concentration of Besifloxacin, Gatifloxacin, and Moxifloxacin in Human Conjunctiva After a Single Topical Instillation
Brief Title: Concentration of Besifloxacin, Gatifloxacin, and Moxifloxacin in Human Conjunctiva After Topical Instillation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 608
Record Dates: First submitted 2009-04-03; First posted 2009-05-21 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: pharmacokinetics
MeSH Terms: interventions — Gatifloxacin; Moxifloxacin; besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Besifloxacin (Experimental): Besifloxacin one drop instilled into study eye.
  Interventions: Drug: Besifloxacin
- Gatifloxacin (Active Comparator): Gatifloxacin one drop instilled into study eye.
  Interventions: Drug: Gatifloxacin
- Moxifloxacin (Active Comparator): Moxifloxacin one drop instilled into study eye.
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Gatifloxacin — Gatifloxacin 0.3% one drop instilled into study eye at visit 2.
  Arms: Gatifloxacin
Drug: Moxifloxacin — Moxifloxacin 0.5% one drop instilled into study eye at visit 2.
  Arms: Moxifloxacin
Drug: Besifloxacin — Besifloxacin 0.6% one drop instilled into study eye at visit 2.
  Other Names: Besivance
  Arms: Besifloxacin

SUMMARY:
The purpose of this study is to assess the concentration of besifloxacin compared to gatifloxacin and moxifloxacin in human conjunctival tissue, following a single drop of the drug instilled topically into the study eye. Conjunctival biopsies will be performed at specified time points, followed by the use of loteprednol etabonate/tobramycin ophthalmic suspension four times a day for 5 days.

ELIGIBILITY:
Inclusion Criteria:

* Willing to avoid all disallowed medications for the appropriate washout periods.
* Have a best corrected visual acuity of 0.60 logMAR or better in each eye as measured using an ETDRS chart.

Exclusion Criteria:

* Have a known allergy and/or sensitivity to the test articles or its components or any therapy associated with the trial.
* Monocular.
* Have previously participated in a conjunctival biopsy study.
* Be currently enrolled in an investigational drug or device study or have uses of an investigational drug or device within 30 days of entry into this study.
* have a condition or is in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Concentration of besifloxacin, gatifloxacin or moxifloxacin in conjunctival tissue. | Biopsies collected at specified time points from 15 minutes to 24 hours

SECONDARY OUTCOMES:
Visual acuity | Day -14 through Day 6(+/-1)
Slit Lamp Biomicroscopy | Day -14 through Day 6 (+/-)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Comstock, OD, Study Director — Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States